CLINICAL TRIAL: NCT04006509
Title: Prenatal Breast Pumping Education of Mothers and Their Support Person
Brief Title: Prenatal Breast Pump Education of Mothers and Their Support Person
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P0081761; IRB201400318 (Other: University of Florida)
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Results first posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Preterm Birth; Breast Feeding
Keywords: preterm breast milk
MeSH Terms: conditions — Premature Birth; Breast Feeding | interventions — Prenatal Education

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antenatal Education Group (Experimental): Patients will receive a prenatally delivered lactation educational program.
  Interventions: Behavioral: Prenatally Delivered Lactation Educational Program
- Standard of Care Group (No Intervention): Patients will receive standard of care and not a prenatally delivered lactation educational program.

INTERVENTIONS:
Behavioral: Prenatally Delivered Lactation Educational Program — The support person (SP) of mothers at risk for preterm birth will be educated on how to use a breast pump and instructions regarding breast milk expression and have a pump in their hospital room
  Other Names: Antenatal Education
  Arms: Antenatal Education Group

SUMMARY:
The study will follow a prospective cohort of racially and economically diverse mothers of premature infants for 3 weeks following delivery to test whether antenatal education of the support person of mothers may decrease time to initiation of breast pumping, decrease time to lactogenesis stage II and increase breast milk production.

DETAILED DESCRIPTION:
Compelling evidence exists that breast milk helps protect premature infants from prematurity-specific morbidities, including feeding intolerance, late onset sepsis, and necrotizing enterocolitis. Unfortunately, mothers of VLBW infants often exhibit delayed lactogenesis stage II (when the milk "comes in") and inadequate breast milk production. Earlier initiation of breast milk expression following delivery is associated with increased lactation success. However, lack of nursing time and lack of hospital personal are significant barriers to the early initiation of milk expression in this population. The proposed study will follow a prospective cohort of racially and economically diverse mothers of premature infants for 3 weeks following delivery to test 1 primary aim and 1 secondary aim. Aim 1: will evaluate the feasibility of antenatal BM pumping education for SPs of mothers of preterm infants. Issues related to recruitment, randomization acceptance of the intervention, and refinement of the education materials and process will be scrutinized. Aim 2 will estimate variability of outcome measurements and effect sizes needed to calculate the sample size for a subsequent larger, adequately powered, randomized clinical trial. Eligible women and their SP will be randomly assigned to one of two groups. Group 1 will receive a prenatally delivered lactation educational program including video recordings, a demonstration of how the pump works and will have a breast pump available in their room. The volume of breast milk produced, timing of lactation stage II, duration of lactation and stress during initial expression will be measured. In addition, breast milk sodium levels will be analyzed on Day 1-7, Day 14 and 21.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* stated intent to breastfeed
* anticipating the birth of a premature infant < 35 weeks gestation.

Exclusion Criteria:

* known illicit maternal drug use
* history of breast reduction or augmentation
* positive HIV status
* infant not expected to live over 2 weeks following delivery.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Parker, Principal Investigator — University of Florida
Locations (1):
- UF Health at the University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker LA, Bendixen M, Sullivan S, Cacho N, Mueller M. Antepartum Breast Pump Education for Mothers and Their Support Person: Effect on Time to First Expression and Lactation Outcomes-A Randomized Controlled Pilot Study. Breastfeed Med. 2022 May;17(5):437-445. doi: 10.1089/bfm.2021.0275. Epub 2022 Apr 26. PMID 35475721

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antenatal Education Group | Standard of Care Group
Started | 49 | 25
Completed | 36 | 25
Not Completed | 13 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antenatal Education Group | Standard of Care Group | Total
Number analyzed (Participants) | 36 | 25 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (6.4) | 29 (6) | 28 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 25 | 61
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 14 | 36
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Onset of Lactogenesis Stage II Through Volume Attainment
Description: Time in hours until mothers pump at least 20 mL of milk in 2 consecutive pumping sessions
Time Frame: Up to 96 Hours
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Antenatal Education Group | Standard of Care Group
Number analyzed (Participants) | 36 | 25
hours | 84.8 [58.8 to 102.6] | 81 [61.3 to 101.3]
Statistical Analysis 1: Comparison: Antenatal Education Group vs Standard of Care Group; Test type: Superiority; p = 0.985, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Breast Milk Production on Day 1
Description: Volume of breast milk produced from 0-24 hours postpartum
Time Frame: 0-24 hours postpartum
Measure: Median (Standard Deviation); unit: mL
Arm/Group | Antenatal Education Group | Standard of Care Group
Number analyzed (Participants) | 36 | 25
mL | 15.3 (16.5) | 24.3 (28.1)
Statistical Analysis 1: Comparison: Antenatal Education Group vs Standard of Care Group; Test type: Superiority; p = 0.539, Marginal Two-Part Model

3. Secondary Outcome: Time to Breast Pumping Initiation
Description: Time to mothers beginning to pump breasts after delivery
Time Frame: first 24 hours after delivery
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Antenatal Education Group | Standard of Care Group
Number analyzed (Participants) | 36 | 25
Hours | 4 (3.5) | 3.8 (3.4)
Statistical Analysis 1: Comparison: Antenatal Education Group vs Standard of Care Group; Test type: Superiority; p = 0.959, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Breast Milk Production Day 2
Description: Volume of breast milk produced on day 2 postpartum
Time Frame: Day 2 postpartum
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Antenatal Education Group | Standard of Care Group
Number analyzed (Participants) | 36 | 25
mL | 32.7 (35.6) | 39.5 (43.7)
Statistical Analysis 1: Comparison: Antenatal Education Group vs Standard of Care Group; Test type: Superiority; p = 0.743, Marginal Two-Part Model

5. Secondary Outcome: Milk Production Day 3
Description: Volume of milk produced on Day 3 postpartum
Time Frame: 3 days postpartum
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Antenatal Education Group | Standard of Care Group
Number analyzed (Participants) | 36 | 24
mL | 55.88 (57.9) | 59.7 (58)
Statistical Analysis 1: Comparison: Antenatal Education Group vs Standard of Care Group; Test type: Superiority; p = 0.886, Marginalized Two-Part Model

6. Secondary Outcome: Breast Milk Production Day 4
Description: Volume of breast milk produced on Day 4 postpartum
Time Frame: Day 4 postpartum
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Antenatal Education Group | Standard of Care Group
Number analyzed (Participants) | 36 | 24
mL | 101.8 (126.6) | 97.4 (87.2)
Statistical Analysis 1: Comparison: Antenatal Education Group vs Standard of Care Group; Test type: Superiority; p = 0.107, Marginalized Two-Part Model

7. Secondary Outcome: Breast Milk Production on Day 5
Description: Volume of breast milk produced on Day 5 postpartum
Time Frame: Day 5 postpartum
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Antenatal Education Group | Standard of Care Group
Number analyzed (Participants) | 36 | 25
mL | 149.9 (167.4) | 138.5 (113.2)
Statistical Analysis 1: Comparison: Antenatal Education Group vs Standard of Care Group; Test type: Superiority; p = 0.687, Marginalized Two-Part Model

8. Secondary Outcome: Breast Milk Production Day 6
Description: Volume of breast milk produced on Day 6 postpartum
Time Frame: Day 6 postpartum
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Antenatal Education Group | Standard of Care Group
Number analyzed (Participants) | 36 | 25
mL | 245.3 (317.9) | 266.8 (300.1)
Statistical Analysis 1: Comparison: Antenatal Education Group vs Standard of Care Group; Test type: Superiority; p = 0.871, Marginalized Two-Part Model

9. Secondary Outcome: Breast Milk Production Day 7
Description: Volume of milk produced on Day 7 postpartum
Time Frame: Day 7 postpartum
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Antenatal Education Group | Standard of Care Group
Number analyzed (Participants) | 36 | 24
mL | 345 (558.4) | 361.9 (342.3)
Statistical Analysis 1: Comparison: Antenatal Education Group vs Standard of Care Group; Test type: Superiority; p = 0.376, Marginalized Two-Part Model

10. Secondary Outcome: Breast Milk Production Day 14
Description: Volume of breast milk produced on Day 14 postpartum
Time Frame: Day 14 postpartum
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Antenatal Education Group | Standard of Care Group
Number analyzed (Participants) | 36 | 25
mL | 431 (416.7) | 428 (349.9)
Statistical Analysis 1: Comparison: Antenatal Education Group vs Standard of Care Group; Test type: Superiority; p = 0.770, Marginalized Two-Part Model

11. Secondary Outcome: Breast Milk Production Day 21
Description: Volume of breast milk produced on Day 21 postpartum
Time Frame: 21 days postpartum
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Antenatal Education Group | Standard of Care Group
Number analyzed (Participants) | 29 | 17
mL | 725 (1070.1) | 573.9 (402.1)
Statistical Analysis 1: Comparison: Antenatal Education Group vs Standard of Care Group; Test type: Superiority; p = 0.237, Marginalized Two-Part Model

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Antenatal Education Group | Standard of Care Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/25
Other Adverse Events (participants affected / at risk) | 0/36 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT04006509/Prot_SAP_000.pdf
  • Informed Consent Form (2011-10-19): https://cdn.clinicaltrials.gov/large-docs/09/NCT04006509/ICF_001.pdf